CLINICAL TRIAL: NCT01288014
Title: Relationship of Cytokine Production and Immune Responses to Varicella Zoster Virus (VZV) in Elderly Recipients of Zoster Vaccine
Brief Title: Cytokine Production and Immunity to Varicella Zoster Virus (VZV) in Elderly Recipients of Zoster Vaccine
Status: Completed | Type: Observational
Sponsor: Columbia University (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Anne A. Gershon, Professor of Pediatrics, Director of the Division of Pediatric Infectious Disease, Columbia University
Other Study IDs: AAAE1779
Record Dates: First submitted 2011-01-31; First posted 2011-02-02 (Estimated); Last update posted 2017-07-19 (Actual); Status verified 2017-07

CONDITIONS: Immunity; Defect Due to Antibody or Cell Mediated Immune Defect
Keywords: immune response; varicella zoster virus (VZV); cytokine levels; immunization
MeSH Terms: conditions — Chickenpox

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Edlerly Recipients of Zoster Vaccine: Blood samples are collected before and after vaccination in people age 60 or more, who are getting the zoster vaccine as part of their routine health care.

SUMMARY:
After immunization, particularly in older persons, some people are protected from disease by a vaccine and others are not. The investigators believe that this variable response may be due to overproduction of molecules that suppress development of immunity (antibodies and cell mediated immunity). Normally, these molecules are produced to make sure that immunity is regulated in just the right way for the body as a whole, and to prevent autoimmune disease.

However, with aging, the immune system may have difficulty in proper immune regulation. Over production of immunosuppressive molecules after vaccination may interfere with the effects of a vaccine. For example when elderly individuals are immunized against zoster with a licensed vaccine, Zostavax, the vaccine is effective in only about 50 to 60%. The investigators will compare blood levels of antibodies, cellular immunity, and immunosuppressive molecules in recipients of Zostavax to see if there is a correlation between development low immunity and high levels of immunosuppressive molecules.

DETAILED DESCRIPTION:
In order to determine whether there is a relationship between production of immunosuppressive cytokines (such as IL-10) an lower levels of immunity to Varicella Zoster Virus (VZV) after vaccination, the investigators will obtain blood samples before and 3-5 times after immunization to determine the immunity to VZV and the levels of certain cytokines. The first blood samples will be obtained before the vaccine is given, as baseline values.

The vaccine being used is the licensed vaccine, Zostavax, which is recommended by the Food and Drug Administration (FDA) and Center for Disease Control and Prevention (CDC) to be administered to all relatively healthy individuals over the age of 50. This study does not concern vaccine safety or effectiveness. As a benefit to vaccines, the vaccine is administered at no charge to the subject.

ELIGIBILITY:
Inclusion Criteria:

* Relatively healthy and over 60 years old

Exclusion Criteria:

* Having already received Zostavax

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Relatively healthy people over age 60 who have not had Zostavax previously.
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2011-01; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Development of antibodies, cellular immunity, and cytokines before and after vaccination | Up to week 6
  Measure antibodies, cellular immunity, and cytokines in blood before and after immunization. Determine if there is any relationship between development of strong immunity and development of cytokine levels.

CONTACTS AND LOCATIONS:
Overall Officials: Anne A. Gershon, MD, Principal Investigator — Columbia University
Locations (1):
- Vanderbilt Clinic, Columbia University Medical Center, New York, New York, United States